CLINICAL TRIAL: NCT00772239
Title: Perioperative Coagulation Management in Cardiac Surgery. Rotem Versus Standard Pratctice. A Randomized Trial.
Brief Title: Perioperative Coagulation Management in Cardiac Surgery.
Acronym: ROTEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Karine Nubret-Le coniat, CHU Limoges
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I07018/ROTEM CTV
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Cardiac Surgery; Bleeding
Keywords: Coagulation Management; Cardiac surgery; Bleeding; Rotem
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotem (Experimental): ROTEM: Rotation thromboelastometry
  Interventions: Device: Rotation thromboelastometry (ROTEM)
- S (Active Comparator): Standard coagulation managment procedure
  Interventions: Procedure: Standard coagulation managment procedure

INTERVENTIONS:
Device: Rotation thromboelastometry (ROTEM) — Coagulation measurement
  Arms: Rotem
Procedure: Standard coagulation managment procedure — Standard coagulation managment procedure
  Arms: S

SUMMARY:
Cardiac surgery is bleeding requiring transfusion surgery .

The haemorrhagic is related to the need to use high doses of anticoagulants to prevent thrombosis of blood . Moreover, this type of surgery is platelets and coagulation factors consumming despite conducting a thorough anticoagulation.

All these changes contribute to increase the need for transfusions during heart surgery.

The main objective of this study is to compare the need for transfusions in patients suffering from bleeding complications after cardiac surgery with a therapeutic algorithm based on the use of ROTEM ® versus standard tests based solely on standard laboratory tests.

100 pateinst (50 in each arm) should be included in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years
* Cardiac surgery or heart transplantation with abnormal bleeding regardless the etiology
* given informed consent

Exclusion Criteria:

* Patient supported by a pre or postoperative circulatory technical assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Quantity of different blood transfusion | during cardiac surgery management

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie NATHAN-DENIZOT, MD, Study Chair — CHU limoges
Locations (4):
- France (4):
  - Service Anésthésie, Limoges, Limoges
  - Service d'Anesthésie, Limoges, Limoges
  - Hôpital Haut Levêque- Service d'Anesthésie réanimation Chirurgicale, Bordeaux
  - Service d'Anesthésie réanimation Chirurgicale, Bordeaux